CLINICAL TRIAL: NCT02350491
Title: Study During Pregnancy of miRNAs in Rheumatoid Arthritis or Systemic Lupus Erythematosus
Brief Title: Study During Pregnancy of Expression of miRNAs in RA or SLE
Acronym: SPIRALE
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 5860
Record Dates: First submitted 2015-01-26; First posted 2015-01-29 (Estimated); Last update posted 2026-02-03 (Actual); Status verified 2017-12

CONDITIONS: Rheumatoid Arthritis; Systemic Lupus Erythematosus
Keywords: Pregnancy; miRNA; Rheumatoid Arthritis (RA); Systemic Lupus Erythematosus (SLE)
MeSH Terms: conditions — Arthritis, Rheumatoid; Lupus Erythematosus, Systemic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The samples that will be analyzed in the present application are serum, urine, placenta, blood monocytes.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- RA group: Pregnant women suffering from Rheumatoid Arthritis.
  Interventions: Other: Collection of biological samples
- SLE group: Pregnant women suffering from Systemic Lupus Erythematosus.
  Interventions: Other: Collection of biological samples
- healthy group: Healthy pregnant woman.
  Interventions: Other: Collection of biological samples

INTERVENTIONS:
Other: Collection of biological samples — collection of biologic samples ( blood and urine) befor and after woman pregnacy

SUMMARY:
Rheumatoid arthritis (RA) is a systemic disease, which mainly targets joints and results in osteoarticular destruction and serious disability. When clinical symptoms (painful and swollen joints) occur, the innate and adaptive immune responses against self antigens have already been largely amplified. This might explain that even when RA patients are treated very early and aggressively, a remission of the disease can only be obtained in approximately half of them. This proportion of remission under treatment can only be achieved using treat to target strategies involving biologics, such as anti-TNF. Unfortunately, less than 20% of patients remain in remission after treatment discontinuation. Thus, despite the availability of 5 different types of biologics, there are still therapeutic unmet needs. However, a spontaneous, drug-free decrease of disease activity can be observed in a physiological condition, pregnancy. Although most of treatments of RA have to be discontinued during pregnancy, a marked improvement, and sometimes remission, can be observed during pregnancy, with frequent post-partum flares. The situation is the opposite with an increased risk of flares in systemic lupus erythematosus (SLE), a rare systemic autoimmune disease which generally progresses in flares-up and can affect nearly any organ (the skin, joints, kidneys, the brain, the heart, …). The course of the disease remains unpredictable for a given patient, and very few biomarkers are available to help clinicians to identify patients a risk of flares. Thus, safe therapeutic options remain limited, especially in patients with serious complications. A specific concern in SLE is the fact that the disease usually starts in women entering their sexual and reproductive life. Even with a stable condition (i.e : lupus without recent flares and no impaired renal or cardiac function) as it is medically recommended before getting pregnant, up to 40% of SLE patients flare up during pregnancy.

We hypothesize disease-specific and pregnancy-induced epigenetic changes, especially those regarding the pattern and levels of microRNAs, could explain the clinical improvement and the risk of flares in RA and SLE, respectively. A better understanding of the underlying mechanisms could help to identify new biomarkers, notably those predicting flares in SLE, and therapeutic targets, by trying to mimicking or amplifying micro-RNA changes observed in RA and targeting them in SLE.

ELIGIBILITY:
Inclusion Criteria:

* ACR criteria for SLE or 2010 ACR criteria for RA
* Absence of any known disease (control group)
* Pregnancy

Exclusion Criteria:

* Age <18
* Other(s) disease(s) that might affect the course of pregnancy (diabetes, uncontrolled hypertension, moderate to severe renal, cardiac or function impairment)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Pregnant women suffering from RA or SLE compared wiht pregnant woman in good health
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-12-17 (Actual); Primary Completion 2018-10-14 (Actual); Study Completion 2018-10-14 (Actual)

PRIMARY OUTCOMES:
To identify the association between pregnancy-induced changes in the pattern of expression of miRNA and disease activity in RA and SLE. | Within the 3 months preceding pregnancy; at diagnosis of pregnancy; after 1 month of pregnancy; after 6 months of pregnancy; at delivery; 1 month after delivery; 3 months after delivery
  The samples that will be analyzed in the present application are serum, urine, placenta, blood monocytes.

CONTACTS AND LOCATIONS:
Overall Officials: Jean SIBILIA, MD, PhD, Study Chair — University Hospital, Strabourg - France; Jacques-Eric GOTTENBERG, Md, PhD, Study Director — niversity Hospital, Strabourg - France
Locations (1):
- Service de rhumatologie Hôpital de Hautepierre, Strasbourg, France

REFERENCES:
- [Result] Scherlinger M, Schmauch E, Carapito R, Pichot A, Alsaleh G, Paul N, Molitor A, Lefebvre F, Schmidt-Mutter C, Bahram S, Sibilia J, Georgel P. Systemic lupus pregnancies are characterized by an intrinsic pro-inflammatory monocyte transcriptome, driven by an aberrant miRNA signature. J Transl Autoimmun. 2025 Dec 24;12:100347. doi: 10.1016/j.jtauto.2025.100347. eCollection 2026 Jun. PMID 41552363